CLINICAL TRIAL: NCT01374230
Title: Long-Term Multicenter Evaluation of the E1® Tibial Bearing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stanford University (Other); Aalborg University Hospital (Other); Göteborg University (Other); Hospital Universitario La Paz (Other); Hvidovre University Hospital (Other); Seoul National University Hospital (Other); Ulsan University Hospital (Other); Sydney Private Hospital, Australia (Unknown); Kennedy Center at Ascension Mercy Hospital (Other); Southern Joint Replacement Institute (Unknown)
Responsible Party: Principal Investigator, Charles R. Bragdon, Associate Director, Clinical Studies, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-001922
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis of the Knee; Traumatic Arthritis of the Knee
Keywords: clinical outcomes; radiographic outcomes; total knee arthroplasty; survivorship
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E1 Tibial bearing (Experimental): All patients undergoing primary total knee replacement surgery will receive a tibial bearing made of E1 polyethylene, which is the material being monitored in this study.
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Primary total knee arthroplasty surgery for the treatment of osteoarthritis.

SUMMARY:
This study has been designed to document the long-term outcome of the E1® Tibial Bearings used with the Vanguard® Knee System in 500 patients receiving total knee arthroplasty. All patients will receive the E1® Tibial Bearing in a Vanguard® knee replacement. Radiographic analysis and patient reported outcomes will be used as follow-up measures to track wear, mechanical performance, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 20 to 75 years of age
* Subjects requiring total knee replacement
* Subjects with the diagnosis of osteoarthritis, or traumatic arthritis
* Subjects who demonstrate the ability to return to Massachusetts General Hospital for follow-up for the next 10 years

Exclusion Criteria:

* Subjects with osteoporosis, osteomalacia, or neuromuscular disease
* Incomplete or insufficient soft tissue around the knee
* Subjects with a limited life span
* Subjects who have difficulty comprehending the study protocol for any reason
* Subjects with disorders which may impair bone formation
* Subjects whose bony structure deviates substantially from the general norm
* Female subjects that are, or may become, pregnant while participating in this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Survivorship, as determined by the implant remaining within the patient. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bragdon, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States